CLINICAL TRIAL: NCT05546879
Title: Study Investigating the Association of NP137 With Atezolizumab-Bevacizumab Combination in First Line in Unresectable Hepatocellular Carcinoma
Brief Title: Study Investigating the Association of NP137 With Atezolizumab-Bevacizumab Combination in First Line in Unresectable HCC
Acronym: Liver-NET1
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Number of patients achieved and treatment ongoing
Sponsor: University Hospital, Grenoble (Other)
Collaborators: NETRIS Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 38RC22.210
Record Dates: First submitted 2022-09-15; First posted 2022-09-21 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — netrin-1 inhibitor NP137; atezolizumab; Bevacizumab

STUDY DESIGN:
Intervention Model Description: Multicentric prospective single arm phase 1b trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): NP137+Atezolizumab-Bevacizumab
  Interventions: Drug: NP137; Drug: Atezolizumab; Drug: Bevacizumab

INTERVENTIONS:
Drug: NP137 — NP137 at 9 or 14 mg/kg IV will be administered every 21 days.
Drug: Atezolizumab — Atezolizumab will be administered by IV infusion at a fixed dose of 1200 mg on Day 1 of each 21-days cycle
Drug: Bevacizumab — Bevacizumab will be administered by IV infusion at a dose of 15 mg/kg on Day 1 of each 21-day cycle

SUMMARY:
The study will assess the safety of the association of NP137 with the standard of care Atezolizumab-Bevacizumab in first line setting in patients with unresectable hepatocellular carcinoma.The study drug which is tested is the NP137 in association with Atezolizumab-Bevacizumab to allow a better tumor response as well as better survival outcomes with an acceptable safety.

DETAILED DESCRIPTION:
The study is a multicentric, prospective, single arm phase 1b trial. This study will enroll 43 to 52 patients and consists of 2 parts: Safety Lead-in Phase and Expansion Phase. Initially, 3 to 12 patients will be enrolled into a Safety Lead-in Phase based on a 3 + 3 design, with the possibility of dose de-escalation, to confirm the recommended dose of NP137 .The Expansion Phase will start after completion of Safety Lead-in Phase at the confirmed dose and will include 40 patients. Patients will be assigned to the experimental single arm (NP137+ Atezolizumab-Bevacizumab).

ELIGIBILITY:
Inclusion Criteria:

1. Males or females ≥ 18 years of age
2. Histologically confirmed (liver biopsy within 24 previous weeks) and documented unresectable hepatocellular carcinoma
3. Patients with a BCLC C or BCLC B status ineligible for or in failure of locoregional treatment, as per the Barcelona Clinic Liver Cancer (BCLC) staging system
4. No prior systemic therapy for advanced HCC
5. Liver tumor burden < 50% of the liver (per Investigator judgment)
6. Child-Pugh A (≤ 6) without any history of cirrhotic decompensation within the past 6 months
7. Antiviral therapy required in hepatitis B virus patients (Hepatitis B antigen positive)
8. Willing to have liver biopsy between C4 and C5
9. Presence of a measurable tumor per RECIST v1.1 criteria
10. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
11. Life expectancy ≥ 12 weeks
12. Absence of previous liver decompensation
13. In case of cirrhosis, last esophageal varices detection by esogastroduodenal endoscopy have to be performed within last the 6 months before inclusion
14. Adequate hematologic function prior to the first dose of NP137, defined as:

    Absolute neutrophils count ≥ 1500 cells/μL 14.2. Hemoglobin ≥ 9 g/dL with no transfusion within 4 weeks prior to first planned dose of NP137 14.3. Platelet count > 50,000/μL with no transfusion within 2 weeks prior to first planned dose of NP137
15. Adequate renal function prior to first dose, defined as:

    15.1. Serum creatinine < 1.5 × Upper limit of normal (ULN ) 15.2. Creatinine clearance ≥ 30 mL/min/m2 (by Cockroft-Gault equation of 24-hour urine) if creatinine ≥ 1.5 × ULN
16. Adequate hepatic function prior first dose, defined as AST/ALT ≤ 5 × ULN
17. Women patients of childbearing potential must have a negative serum pregnancy test at screening and baseline, and be willing to use a highly effective contraception. The patient should be advised to continue the contraception for at least 6 months following the completion of dosing. Women with cessation for > 24 months of previously occurring menses, or women of any age who have had a hysterectomy, or have had both ovaries removed will be considered to be of non-childbearing potential.
18. Male patients of reproductive potential must be willing to use one acceptable method of contraception, as judged by Investigator and Sponsor and/or to refrain from donating sperm from the time of screening through at least 6 months following the completion of dose administration.
19. Amenable to computed tomography (CT) with 3 or 4 phase liver or magnetic resonance imaging (MRI) of abdomen and pelvis, and CT of chest, or MRI of whole body, for initial tumor size measurements and subsequent follow-up.
20. Absence of other clinically relevant abnormalities for any screening laboratory test results as judged by the Investigator and Sponsor.
21. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
22. Able to understand and provide written informed consent
23. Patients covered by Health Insurance System

Exclusion Criteria:

1. Any known history of encephalopathy within 6 months prior to first planned dose of treatment
2. Untreated or incompletely treated esophageal and/or gastric varices with bleeding or high-risk for bleeding
3. Known esophageal varices with recent history of bleeding (within previous 6 months)
4. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures
5. Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC
6. Chronic treatment with immunosuppressive agents (like steroids) ≤ 6 weeks prior to first planned dose of treatment.
7. Major surgical procedures, open biopsy or significant traumatic injury ≤ 4 weeks prior to first dose of treatment or anticipation of major surgical procedure during the course of the trial, minor surgical procedures ≤ 1 week of first planned dose (the surgical wound must be fully healed)
8. Local therapy to liver within 28 days prior to initiation of study treatment or non-recovery from side effects of any such procedure
9. Any clinically significant cardiovascular condition as judged by the Investigator (such as New York Heart Association Class II or greater cardiac failure, myocardial infarction, or cerebrovascular accident within 3 months prior to Day 1 of Cycle 1, uncontrolled arterial hypertension, unstable arrhythmia, or unstable angina)
10. Severe or uncontrolled renal condition
11. Untreated chronic hepatitis B
12. Co-infection of HBV and HCV
13. Use of any prohibited concomitant medications within 14 days of the Baseline/Day 1 visit
14. Contraindication to additionnal liver biopsy planned between C4 and C5
15. Contraindication to iodinated contrast agent infusion
16. Known current alcohol (> 20g/ Day in women and > 30g/ Day in men) or substance abuse
17. History of leptomeningeal disease
18. Active or history of autoimmune disease or immune deficiency
19. History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography scan
20. Known active tuberculosis
21. History of malignancy other than HCC within 5 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death
22. Pregnancy or breastfeeding, or intention of becoming pregnant during study treatment or within at least 6 months after the last dose of treatment
23. Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases
24. Uncontrolled tumor-related pain
25. Uncontrolled or symptomatic hypercalcemia
26. Treatment with systemic immunostimulatory agents
27. Inadequately controlled arterial hypertension
28. Prior history of hypertensive crisis or hypertensive encephalopathy
29. Evidence of bleeding diathesis or significant coagulopathy
30. History of intestinal obstruction and/or clinical signs or symptoms of GI obstruction including sub-occlusive disease related to the underlying disease or requirement for routine parenteral hydration
31. Serious, non-healing or dehiscing wound, active ulcer, or untreated bone fracture
32. Metastatic disease that involves major airways or blood vessels, or centrally located mediastinal tumor masses
33. Known clinically significant or life threatening organ or systemic disease such that in the opinion of the Investigator, the significance of the disease will compromise the patient's participation in the trial
34. Known intolerance or hypersensitivity to the active ingredient or to one of the components of the study drug
35. Persistent toxicities related to prior treatment of grade greater than 1
36. Subjects with active infection
37. History of bone marrow allograft or solid organ transplant
38. Subjects requiring corticosteroid therapy at a dose equivalent to more than 10 mg of prednisone equivalent dose per day (corticosteroid administration is permitted by a route resulting in minimal systemic exposure [cutaneous, rectal, articular, ocular or inhalation] is authorized).
39. Hypersensitivity to Chinese Hamster Ovary (CHO) cell products or other recombinant human or humanised antibodies
40. History of gastrointestinal perforations and fistulae
41. Uncontrolled or symptomatic proteinuria
42. Active aneurysm considered as unstable and/or at high risk of complication
43. Patients who experienced immune-mediated pericardial disorders during previous treatment by immune checkpoint blockade therapies, including anti-CTLA4, anti-PD1, and anti-PDL1 therapeutic antibodies
44. Subject who participate or plan to participate in another interventional clinical trial or who is in exclusion period for another study,
45. Subject who cannot be contacted in case of emergency
46. Persons referred to in Articles L1121-5 to L1121-8 of the French code of public health (this corresponds to all persons protected: pregnant or parturient women, breastfeeding mothers, persons deprived of liberty by judicial or administrative decision, persons subject to a legal protection measure).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
Percentage Proportion of patients experiencing adverse events | At 36 months
  Percentage Proportion of patients experiencing adverse events (AEs) of any grade and grade 3/4 AEs as defined by the National Cancer Institute - Common Terminology Criteria for Adverse Events (CTCAE v 5.0) throughout the study period.

SECONDARY OUTCOMES:
Best overall objective response rate (ORR) | At 36 months
  Best overall objective response rate (ORR) and ORR at 3 months, 6, 9, 12 months according to mRECIST and RECIST 1.1.
Overall survival (OS) | At 36 months
  Median Overall survival (OS) at 6 months- and 12 months-OS rates. OS is defined as the time between inclusion and death (all causes). Patients alive will be censored at the date of last news.
Progression-Free Survival (PFS) | At 36 months
  Median Progression-Free Survival (PFS) at 6 months- and 12 months-PFS rates according to RECIST 1.1.
Duration of response | At 36 months
  Median Duration of response is defined as the time between first dose of treatment and progression according to RECIST 1.1. Patients alive without progression will be censored at 6 months and at the date of last news.
Alpha-fetoprotein (AFP) response | At 36 months
  AFP response will be defined as a percentage of patients with a ≥ 50% reduction from baseline AFP level, at 3, 6, 12 months
Quality of life (QoL) | At 36 months
  QoL will be studied by using the European Organisation for Research and Treatment of Cancer Quality-of-Life Questionnaire for Cancer at baseline, 3, 6, 12 months. A 5-point decrease of QLQ-C30 score will be considered as the minimal clinically significant deterioration of QoL.
time to deterioration (TTD) | At 36 months
  TTD will be defined as the time from inclusion in the study to deterioration of EORTC QLQ-C30 score with a decrease ≥5 points at any time point after the baseline score at 6 months and at the end of study.
PK-PD evaluation | At 36 months
  based on available PopPK modelisation and PK samples collected at the time of the response evaluation in this study
Mechanism of EMT | At 36 months
  To assess the mechanisms of EMT reversal by comparing different histological markers on pre-therapeutic and Cycle4-Cycle5 biopsies. Descriptive study in transcriptomics and immunohistochemistry of the evolution of EMT markers, Netrin-1 expression, and tumor microenvironment during treatment by comparing pre-therapeutic biopsies to Cycle4-Cycle5 biopsies

CONTACTS AND LOCATIONS:
Overall Officials: Gaël ROTH, MD PHD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- CHU de GRENOBLE ALPES, Grenoble, Alpes, France

IPD SHARING:
Plan to Share IPD: No